CLINICAL TRIAL: NCT07055672
Title: Clinical Effectiveness of the Modified WalkFlex DB Splint in Children With Congenital Talipes Equinovarus (CTEV): A Prospective Pilot Study.
Brief Title: Clinical Effectiveness of the Modified WalkFlex DB Splint in Children With Congenital Talipes Equinovarus (CTEV)
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: MSRSW/Batch-Fall23/827
Record Dates: First submitted 2025-06-28; First posted 2025-07-09 (Actual); Last update posted 2025-07-09 (Actual); Status verified 2025-06

CONDITIONS: Congenital Talipes Equinovarus
MeSH Terms: conditions — Clubfoot

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Combination Product: Modified WalkFlex DB Splint (Intervention Arm) — Application of the Modified WalkFlex Denis Browne (DB) Splint
  Children with corrected idiopathic clubfoot will use the Modified WalkFlex DB Splint for maintenance. This splint allows knee and some hip movement and includes a detachable bar for walking. It will be used after Ponseti casting, and patients will be followed at 1 and 3 months to check splint tolerance, maintenance of correction (using Pirani score), and any signs of relapse

SUMMARY:
This pilot study aims to evaluate the effectiveness of the Modified WalkFlex DB Splint in the maintenance phase of Congenital Talipes Equinovarus (CTEV) treatment following successful correction through the Ponseti method. The traditional Denis Browne splint, though widely used, often limits patient mobility and can result in poor compliance. In response to these limitations, the Modified WalkFlex DB Splint was designed to offer increased flexibility at the knee and hip joints, allowing for improved function and easier ambulation while maintaining foot correction.

DETAILED DESCRIPTION:
This is a prospective observational study including 12-15 children aged between 3 months to 3 years who have completed the casting phase.

ELIGIBILITY:
Inclusion Criteria:

* children aged 3 months to 3 years diagnosed with idiopathic congenital talipes equinovarus (CTEV)
* who have completed the correction phase using the Ponseti method and are starting the bracing phase.
* Informed consent from parents or guardians and willingness to attend follow-ups at 1 and 3 months is required

Exclusion Criteria:

* Children with non-idiopathic clubfoot (e.g., syndromic or neuromuscular)
* other congenital limb deformities
* or poor compliance with treatment and follow-up will be excluded

Ages: 3 Months to 3 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 15 (Actual)
Dates: Start 2025-03-17 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Pirani Score | 12 Months
  Used to assess the severity of clubfoot deformity. It consists of six clinical signs divided into midfoot and hindfoot scores. Each sign is scored as 0 (normal), 0.5 (moderate), or 1 (severe). The total score ranges from 0 (normal foot) to 6 (severe deformity).
Relapse Assessment Checklist (Clinical Observation) | 12 Months
  Observation-based checklist used at 1-month and 3-month follow-ups to check for signs of relapse such as equinus, varus, adductus, or cavus. Relapse is defined as the recurrence of one or more of these deformities after initial correction.
Parental/Guardian Feedback Questionnaire (Custom/Adapted) | 12 Months
  A structured feedback form to assess splint tolerance, ease of use, and parental satisfaction. Responses are collected using a 5-point Likert scale (1 = Strongly Disagree, 5 = Strongly Agree) on questions regarding comfort, usability, and perceived effectiveness of the splint.

CONTACTS AND LOCATIONS:
Locations (1):
- Ghurki trust and teaching hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No